CLINICAL TRIAL: NCT01283750
Title: Maximizing Independence at Home (MIND at Home): Dementia Care at Home Study
Brief Title: Maximizing Independence at Home (MIND at Home)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Jewish Community Federation of Baltimore (Unknown); Jewish Community Services (Other); Levindale (Unknown); The Harry & Jeanette Weinberg Foundation, Inc. (Other); Leonard & Helen R. Stulman Charitable Foundation (Unknown); Hoffberger Foundation (Unknown); Hirschhorn Foundation (Other); Lois and Irving Blum Foundation (Unknown); Joseph and Harvey Meyerhoff Family Charitable Funds (Unknown); The Henry and Ruth Blaustein Rosenberg Foundation (Unknown); Baltimore County Department of Aging (Unknown); National Institute of Mental Health (NIMH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00012829; 90032824 (Other: Other)
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Memory Disorders; Dementia
Keywords: care coordination; dementia care; intervention; unmet needs; community; older adults; caregiver
MeSH Terms: conditions — Memory Disorders; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Augmented Usual Care (No Intervention)
  Interventions: Behavioral: care coordination

INTERVENTIONS:
Behavioral: care coordination — dementia-related care coordination

SUMMARY:
Funded by a unique private philanthropy and public coalition through THE ASSOCIATED: Jewish Community Federation of Baltimore, this project seeks to develop effective ways to deliver dementia care to older adults with memory disorders who live in the community. MIND at Home is an 18 month intervention research study whose goals are two-fold: To partner with community organizations to help proactively identify older adults in the Baltimore community who may need help related to memory disorders; To find out if providing person-centered, coordinated care will help older adults with memory disorders remain at home longer, as well other possible benefits. The investigators hypothesize that individuals with memory disorders that receive person-centered, coordinated care will have fewer unmet dementia-related needs, improved quality of life and function, fewer behavioral and depressive symptoms, and will be able to remain in their homes longer compared to individuals who receive augmented usual care.

ELIGIBILITY:
Inclusion Criteria:

* 70+ years old
* Community living (within one of 28 zip codes in Baltimore)
* Has memory disorder
* Has identified study partner willing to participate
* English-speaking

Exclusion Criteria:

* Situation at the time of referral is an emergency with risk of danger to individual or others
* Presence of delirium or other rule outs for memory disorder

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 303 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in unmet dementia-related needs from Baseline to 18 months | 18 months
  Unmet dementia-related needs as measured by the Johns Hopkins Dementia Care Needs Assessment (JHDCNA), clinican-based assessment of 21 domains (92 individual items)

SECONDARY OUTCOMES:
Change in quality of life from Baseline to 18 months | 18 month
  Participant quality of life measured by Quality of Life in Alzheimers Disease (QOL-AD) and Alzheimer's Disease Related Quality of life scale (ADRQL). Caregiver quality of life measured by SF-12.
length of stay | 18 months
  Length of stay in the community assessed by number of days from initial study assessment to end of study observation or to date that the subject leaves their community-based residence (e.g. move to nursing home, assisted living, death) prior to end of study observation.
neuropsychiatric behavior symptoms from baseline to 18 months | 18 month
  Neuropsychiatric behavior measured by the Neuropsychiatry Inventory Questionnaire
day-to-day function from baseline to 18 months | 18 month
  Day-to-day function assessed by the Instrumental Activities of Daily Living Scale and the Psycho-geriatric Dependency Rating Scale
health care utilization from baseline to 18 months | 18 month
  Inpatient, residential, Alzheimer Disease-related, mental health, and medical health care use measured by the SURFS
depression from baseline to 18 months | 18 month
  Participant depression measured by the Cornell Scale for Depression (CSDD) in Dementia. Caregiver depression measured by the Geriatric Depression Scale (GDS).

CONTACTS AND LOCATIONS:
Overall Officials: Quincy M Samus, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Johnston D, Samus QM, Morrison A, Leoutsakos JS, Hicks K, Handel S, Rye R, Robbins B, Rabins PV, Lyketsos CG, Black BS. Identification of community-residing individuals with dementia and their unmet needs for care. Int J Geriatr Psychiatry. 2011 Mar;26(3):292-8. doi: 10.1002/gps.2527. Epub 2010 Jul 23. PMID 20658473
- [Result] Marquardt G, Johnston D, Black BS, Morrison A, Rosenblatt A, Lyketsos CG, Samus QM. Association of the spatial layout of the home and ADL abilities among older adults with dementia. Am J Alzheimers Dis Other Demen. 2011 Feb;26(1):51-7. doi: 10.1177/1533317510387584. PMID 21282278
- [Result] Marquardt G, Johnston D, Black BS, Morrison A, Rosenblatt A, Lyketsos CG, Samus QM. A Descriptive Study of Home Modifications for People with Dementia and Barriers to Implementation. J Hous Elderly. 2011 Jan 1;25(3):258-273. doi: 10.1080/02763893.2011.595612. PMID 21904419
- [Result] Black BS, Johnston D, Morrison A, Rabins PV, Lyketsos CG, Samus QM. Quality of life of community-residing persons with dementia based on self-rated and caregiver-rated measures. Qual Life Res. 2012 Oct;21(8):1379-89. doi: 10.1007/s11136-011-0044-z. Epub 2011 Oct 26. PMID 22038392
- [Result] Samus QM, Johnston D, Black BS, Hess E, Lyman C, Vavilikolanu A, Pollutra J, Leoutsakos JM, Gitlin LN, Rabins PV, Lyketsos CG. A multidimensional home-based care coordination intervention for elders with memory disorders: the maximizing independence at home (MIND) pilot randomized trial. Am J Geriatr Psychiatry. 2014 Apr;22(4):398-414. doi: 10.1016/j.jagp.2013.12.175. Epub 2014 Jan 4. PMID 24502822
- [Result] Black BS, Johnston D, Rabins PV, Morrison A, Lyketsos C, Samus QM. Unmet needs of community-residing persons with dementia and their informal caregivers: findings from the maximizing independence at home study. J Am Geriatr Soc. 2013 Dec;61(12):2087-2095. doi: 10.1111/jgs.12549. PMID 24479141
- See also: Johns Hopkins University press release (2/10/14) — http://www.hopkinsmedicine.org/news/media/releases/experimental_care_program_keeps_people_with_dementia_at_home_longer_study_shows